CLINICAL TRIAL: NCT02362230
Title: Sun Yat-sen University Cancer Center
Brief Title: Evaluation of Icotinib in Metastatic Triple-negative Breast Cancer After Second-line Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty accruing subjects the study accrual was closed
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-006
Record Dates: First submitted 2015-02-08; First posted 2015-02-12 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib (Experimental): Icotinib 125 mg BID
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Icotinib 125 mg BID
  Other Names: Conmana

SUMMARY:
Evaluating the safety and efficacy of Icotinib administered in 2-month treatments, in patients with metastatic triple-negative breast cancer that have received at least two prior treatments.

DETAILED DESCRIPTION:
This is a phase II, multi-center study. Sixty-seven patients are planned to be enrolled. All patients will receive Icotinib 125 mg BID administered for 8 weeks. Patients with a complete response, partial response or stable disease at that time may continue to be treated based on physician discretion. Follow up is then required until resolution or stabilization of any treatment-related toxicity, and patients with stable disease or objective responses must also continue evaluations until survived.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* ECOG 0 or 1
* Primary or metastatic tumor onfirmed as triple negative
* Measurable disease per RECIST version 1.1
* normal organ function, including bone marrow function, renal function, liver function, and cardiac function
* Two or more prior chemotherapy
* signed and dated an informed consent form
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Pregnant or breast feeding
* ECOG score ≧2
* Uncontrolled medical problems
* Hepatic, renal, or bone marrow dysfunction as detailed above
* Concurrent malignancy or history of other malignancy within the last five years except as noted above
* Patients were unable or unwilling to comply with program requirements

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 36 months
  the time from randomization to the date of disease progression or death from any causes

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-Yu Yuan, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No